CLINICAL TRIAL: NCT02221648
Title: Investigation of Efficacy of Botulinum Toxin A (Dysport) in Chronic Low Back Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI retired and moved- funding sponsor contacted and Oked
Sponsor: Yale University (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1210011010
Record Dates: First submitted 2014-04-01; First posted 2014-08-20 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lower Back Pain
Keywords: Back; Pain; Muscle
MeSH Terms: conditions — Low Back Pain; Pain | interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomization to receive injections with either the study drug (abobotulinumtoxinA) or the placebo group. The subjects will be blinded to which intervention they will receive.
  Interventions: Drug: Placebo
- AbobotulinumtoxinA Treatment (Active Comparator): Subjects will be randomized to receive intervention injections with the study drug arbobotulinumtoxinA.
  Interventions: Drug: AbobotulinumtoxinA Treatment

INTERVENTIONS:
Drug: Placebo — Subjects will be randomization to receive either the study drug or the placebo group.
  Arms: Placebo
Drug: AbobotulinumtoxinA Treatment — Subjects receive intervention injections with the study drug arbobotulinumtoxinA.
  Other Names: Dysport
  Arms: AbobotulinumtoxinA Treatment

SUMMARY:
The scientific aim of this study is to investigate the efficacy of abobotulinumtoxinA (Dysport - Ipsen Pharmaceuticals) in chronic low back pain.

The investigators hypothesis is that injection of Dysport brand of botulinum toxin type A into erector spinae muscles (extensors of the spine) can relieve low back pain through anti-spasm and analgesic effect of botulinum toxin.

DETAILED DESCRIPTION:
This is an investigator initiated, randomized, double blind, placebo-controlled study. A total of 90 patients will be enrolled in the study. The study will be conducted over 4 months. It includes 4 visits and 4 telephone calls. Patients with chronic low back pain (>3 months) who meet inclusion and exclusion criteria and wish to participate in the study may be enrolled. Those who become enrolled will be scheduled for a baseline visit (Week 0). During the baseline visit, subjects will be given the official approved consent form to read and ask questions. Participants to this study will also receive a copy of the Dysport Risk Evaluation and Mitigation Strategy (REMS) statement. After obtaining informed consent signed by the subject, the subjects will be randomization into the Dysport or placebo group. The randomizing will be performed by a nurse and the information will be kept in a pass-worded computer. Blinding means that neither the participant nor the clinical rater will know which group the participant has been initially been assigned.

Each subject will have a neurological examination and fill a demographic form and complete four rating questionnaires (appendix II-V). These include a visual analogue scale for pain (0 to 10) and three quality of life questionnaires which depict quality of life (the American Chronic Pain Association's Quality of Life Scale), how pain affects ability to manage everyday life (Oswestry Low Back Pain Disability Questionnaire), and overall physical and emotional health (Short Form-36). Patients will then receive an injection of either abobotulinumA (Dysport) or normal saline. Dysport or saline will be administered into the paraspinal muscles (extensors or erector spinae) at five levels (L1-L5), regardless of pain location. In the case of unilateral pain, this would amount to 500 units total, and in the case of bilateral pain, to 1000 units total, of Dysport per session.

The primary outcome of the study is number of patients with VAS < 4 ( no or subtle pain) at week 6 after placebo or Dysport injection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80, all ethnic groups, races, both sexes.
* Diagnosis of chronic low back pain (longer than 3 months).
* Pain of moderate to severe intensity (VAS 4 or higher).
* Subjects who are able to read, speak, and understand English.

Exclusion Criteria:

Existing significant acute medical condition (i.e. cardiovascular, endocrine, hematologic, neoplastic, infectious, or autoimmune disorders).

* Hypersensitivity to any botulinum toxin product or is recipient
* Allergy to albumin. Lactose or cow milk protein
* Infection in the proposed injection site.
* Pregnancy or planned pregnancy (determined by urine pregnancy test). The women of childbearing age should use a reliable mode of contraception during the study period (abstinence, etc).
* Active breast feeding.
* Enrollment in any clinical trial (currently or within the past 3 months) in which treatments are imposed by a protocol.
* Patients taking high doses of aminoglycosides or other drugs affecting the function of neuromuscular junction (anticholinergics , muscle relaxants)
* Subjects who are younger than 18 years of age.
* Neuromuscular-junction disorders and motor neuron disease such as Amyotrophic Lateral Sclerosis.
* Evidence of acute pathology on neuro-imaging.
* Axis I diagnosis determined by a neurologist or psychiatrist.
* Anesthetic medications within two weeks and corticosteroid injections within 4 weeks of enrollment.
* Received botulinum toxin injections in the past 3 months.
* History of low back surgery , evidence of acute disc or severe lumbar stenosis in MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Jabbari, MD, Principal Investigator — Yale University
Locations (1):
- Yale Medical Group, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to relocation of PI, study was terminated with 43 enrollments(total).
Groups:
- Placebo: Subjects will be randomized to receive injections with either the study drug (abobotulinumtoxinA) or the placebo group. The subjects will be blinded to which intervention they will receive for the first injections.
- ArbobotulinumtoxinA Treatment: Subjects will receive intervention injections with the study drug abobotulinumtoxinA.
  AbobotulinumtoxinA Treatment: All subjects will receive intervention injections with the study drug arbobotulinumtoxinA. A series of rating scale and an examination will take place prior to treatment and at 4 and 8 weeks post treatment.
Period: Overall Study
Arm/Group | Placebo | ArbobotulinumtoxinA Treatment
Started | 22 | 21
Completed | 19 | 18
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects will be randomization to receive injections with either the study drug (incobotulinumtoxinA) or the placebo group. The subjects will be blinded to which intervention they will receive for the first injections.
- AbobotulinumtoxinA Treatment: All subjects will receive intervention injections with the study drug abobotulinumtoxinA.
- Total: Total of all reporting groups
Arm/Group | Placebo | AbobotulinumtoxinA Treatment | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Mild or no Pain on Visual Analog Scale (VAS)
Description: The primary outcome measure in this protocol is the proportion of subjects that have VAS <4 (patients with no or mild pain) at week 6. The pain VAS is a continuous scale comprised of a line 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10).
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Placebo: Subjects will be randomized to receive injections with saline.
- AbobotulinumtoxinA Treatment: All subjects will receive intervention injections with the study drug arbobotulinumtoxinA.
Arm/Group | Placebo | AbobotulinumtoxinA Treatment
Number analyzed (Participants) | 19 | 18
participants | 3 | 5
Statistical Analysis 1: Comparison: Placebo vs AbobotulinumtoxinA Treatment; Test type: Superiority or Other; p = 0.4470, Fisher Exact

2. Secondary Outcome: Number of Patients With Improved Pain Using the Patient Global Impression of Change (PGIC)
Description: The PGIC is a 7 point scale that requires the clinician to assess how much the patient's pain has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:
  No change (or condition has gotten worse) (1) Almost the same, hardly any change at all (2) A little better, but no noticeable change (3) Somewhat better, but the change has not made any real difference (4) Moderately better, and a slight but noticeable change (5) Better and a definite improvement that has made a real and worthwhile difference (6) A great deal better and a considerable improvement that has made all the difference (7)
  This outcome is number of patients who chose a 6 or above on the PGIC 6 weeks after treatment
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Placebo: Study group received placebo injection.
- botulinumtoxinA Treatment: Subjects received botox injection.
Arm/Group | Placebo | botulinumtoxinA Treatment
Number analyzed (Participants) | 19 | 18
participants | 2 | 8
Statistical Analysis 1: Comparison: Placebo vs botulinumtoxinA Treatment; Test type: Superiority or Other; p = 0.0293, Fisher Exact

3. Secondary Outcome: Number of Subjects Showing Improvement on Quality of Life Scale for Pain
Description: The Quality of Life Scale: A Measure of Function for People With Pain was developed by the American Chronic Pain Association (ACPA). The patient is asked to rank their quality of life on a scale of zero (non-functioning) to 10 (normal quality of life). Improvement was defined as 2 or more grades of improvement on the scale.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | AbobotulinumtoxinA Treatment
Number analyzed (Participants) | 19 | 18
participants | 4 | 10
Statistical Analysis 1: Comparison: Placebo vs AbobotulinumtoxinA Treatment; Test type: Superiority or Other; p = 0.0448, Fisher Exact

ADVERSE EVENTS:
Groups:
- Placebo: Subjects will be randomized to receive injections with placebo.
- ArbobotulinumtoxinA Treatment: AbobotulinumtoxinA Treatment: All subjects will receive intervention injections with the study drug arbobotulinumtoxinA.
Arm/Group | Placebo | ArbobotulinumtoxinA Treatment
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

LIMITATIONS AND CAVEATS:
This study was terminated due to relocation of the PI. The initial goal was enrolling 90 patients. The number enrolled at the time of termination was 43, with 37 completed the study. Results may not provide enough statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No